CLINICAL TRIAL: NCT03424005
Title: A Phase Ib/II, Open-label, Multicenter, Randomized Umbrella Study Evaluating the Efficacy and Safety of Multiple Treatment Combinations in Patients With Metastatic Breast Cancer (Morpheus-panBC)
Brief Title: A Study Evaluating the Efficacy and Safety of Multiple Treatment Combinations in Patients With Metastatic or Locally Advanced Breast Cancer
Acronym: Morpheus-panBC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Gilead Sciences (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO40115; 2017-002038-21 (EudraCT Number); 2023-503629-20-00 (EU CTIS Number)
Record Dates: First submitted 2018-01-30; First posted 2018-02-06 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; atezolizumab; ipatasertib; SGN-LIV1A; Bevacizumab; Drug Therapy; Gemcitabine; Carboplatin; eribulin; selicrelumab; tocilizumab; 130-nm albumin-bound paclitaxel; sacituzumab govitecan; abemaciclib; Fulvestrant; ribociclib; inavolisib; trastuzumab deruxtecan; Letrozole; empagliflozin; palbociclib; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (19):
- Atezolizumab + Nab-Paclitaxel (Active Comparator): 1L PD-L1-positive participants will receive doublet combination treatment with atezolizumab plus nab-paclitaxel until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Enrollment is closed.
  Interventions: Drug: Atezolizumab; Drug: Nab-Paclitaxel
- Atezolizumab + Nab-Paclitaxel + Tocilizumab (Experimental): 1L PD-L1-positive participants will receive combination treatment with atezolizumab plus nab-paclitaxel and tocilizumab until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Enrollment is closed.
  Interventions: Drug: Atezolizumab; Drug: Tocilizumab; Drug: Nab-Paclitaxel
- Atezolizumab + Sacituzumab Govitecan (Experimental): 1L PD-L1-positive participants will receive doublet combination treatment with atezolizumab plus sacituzumab govitecan until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Enrollment is closed.
  Interventions: Drug: Atezolizumab; Drug: Sacituzumab Govitecan
- Capecitabine (Active Comparator): 2L CIT-naïve participants will receive capecitabine until unacceptable toxicity or disease progression per Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1).
  Participants who progressed on treatment may have the option of receiving atezolizumab along with chemotherapy (chemo) during stage 2, provided they meet the eligibility criteria.
  Enrollment is closed.
  Interventions: Drug: Capecitabine
- Atezolizumab + Ipatasertib (Experimental): 2L CIT-naïve participants will receive doublet combination treatment with atezolizumab plus ipatasertib until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Participants who progressed on treatment may have the option of receiving atezolizumab + chemo, provided they meet the eligibility criteria.
  Enrollment is closed and participant follow-up is complete.
  Interventions: Drug: Atezolizumab; Drug: Ipatasertib
- Atezolizumab + SGN-LIV1A (Experimental): 2L CIT-naïve participants will receive doublet combination treatment with atezolizumab plus SGNLIV1A until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Patients who experience loss of clinical benefit as determined by the investigator or unacceptable toxicity related to SGN-LIV1A will be given the option of receiving Atezolizumab + chemo during Stage 2, provided they meet the eligibility criteria.
  Enrollment is closed.
  Interventions: Drug: Atezolizumab; Drug: SGN-LIV1A
- Atezolizumab + Selicrelumab + Bevacizumab (Experimental): 2L-CIT-naïve participants will receive doublet combination treatment with atezolizumab plus selicrelumab and bevacizumab until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Participants who progressed on treatment may have the option of receiving atezolizumab + chemo, provided they meet the eligibility criteria.
  Enrollment is closed and participant follow-up is complete.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Selicrelumab
- Atezolizumab + Chemo (Gemcitabine + Carboplatin or Eribulin) (Experimental): 2L CIT-naïve participants enrolled in the active comparator arm who experience disease progression per RECIST v1.1 and 2L CIT-naïve participants enrolled in an experimental arm who experience loss of clinical benefit as determined by the investigator may receive doublet combination treatment with atezolizumab plus chemo (gemcitabine + carboplatin or eribulin) until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Enrollment is closed and participant follow-up is complete.
  Interventions: Drug: Atezolizumab; Drug: Chemotherapy (Gemcitabine + Carboplatin or Eribulin)
- Inavolisib + Abemaciclib + Fulvestrant (Experimental): HR+ participants will receive treatment with inavolisib plus abemaciclib plus fulvestrant until unacceptable toxicity or disease progression determined by the investigator according to RECIST v1.1.
  Interventions: Drug: Abemaciclib; Drug: Fulvestrant; Drug: Inavolisib
- Inavolisib + Ribociclib (Dose #1) + Fulvestrant (Experimental): HR+ participants will receive treatment with inavolisib plus ribociclib plus fulvestrant until unacceptable toxicity or disease progression as determined by the investigator according to RECIST v1.1.
  Interventions: Drug: Fulvestrant; Drug: Ribociclib (Dose #1); Drug: Inavolisib
- Inavolisib + Ribociclib (Dose #1) + Letrozole (Experimental): HR+ participants will receive treatment with inavolisib plus ribociclib plus letrozole until unacceptable toxicity or disease progression as determined by the investigator according to RECIST v1.1.
  Interventions: Drug: Ribociclib (Dose #1); Drug: Letrozole; Drug: Inavolisib
- Inavolisib + Ribociclib (Dose #2) + Fulvestrant (Experimental): HR+ participants will receive treatment with inavolisib plus ribociclib plus fulvestrant until unacceptable toxicity or disease progression as determined by the investigator according to RECIST v1.1.
  Interventions: Drug: Fulvestrant; Drug: Ribociclib (Dose #2); Drug: Inavolisib
- Inavolisib + Ribociclib (Dose #2) + Letrozole (Experimental): HR+ participants will receive treatment with inavolisib plus ribociclib plus letrozole until unacceptable toxicity or disease progression as determined by the investigator according to RECIST v1.1.
  Interventions: Drug: Ribociclib (Dose #2); Drug: Letrozole; Drug: Inavolisib
- Inavolisib + Abemaciclib + Letrozole (Experimental): HR+ participants will receive treatment with inavolisib plus abemaciclib plus letrozole until unacceptable toxicity or disease progression as determined by the investigator according to RECIST v1.1.
  Interventions: Drug: Abemaciclib; Drug: Letrozole; Drug: Inavolisib
- Inavolisib (Dose #1) + Trastuzumab Deruxtecan (Experimental): HER2+/HER2-low participants will receive inavolisib + trastuzumab deruxtecan until unacceptable toxicity or disease progression as determined by the investigator according to RECIST v1.1.
  Interventions: Drug: Inavolisib (Dose #1); Drug: Trastuzumab Deruxtecan
- Inavolisib (Dose #2) + Trastuzumab Deruxtecan (Experimental): HER2+/HER2-low participants will receive inavolisib + trastuzumab deruxtecan until unacceptable toxicity or disease progression as determined by the investigator according to RECIST v1.1.
  Interventions: Drug: Trastuzumab Deruxtecan; Drug: Inavolisib (Dose #2)
- Empagliflozin (Empa) + Inavolisib (Inavo) + Fulvestrant (Fulv) ± Palbociclib (Palbo) (Experimental): Participants with locally advanced or metastatic, HR+, HER2- participants will receive empagliflozin plus inavolisib plus fulvestrant with or without palbociclib until unacceptable toxicity or disease progression as determined by the investigator according to RECIST v1.1.
  Interventions: Drug: Fulvestrant; Drug: Inavolisib; Drug: Empagliflozin; Drug: Palbociclib
- Metformin (Metf) + Inavolisib + Fulvestrant ± Palbociclib (Experimental): Participants with locally advanced or metastatic, HR+, HER2- participants will receive metformin plus inavolisib plus fulvestrant with or without palbociclib until unacceptable toxicity or disease progression as determined by the investigator according to RECIST v1.1.
  Interventions: Drug: Fulvestrant; Drug: Inavolisib; Drug: Palbociclib; Drug: Metformin
- Inavolisib + Atirmociclib (Atirmo) + Fulvestrant (Experimental): Participants will receive inavolisib plus atirmociclib plus fulvestrant until unacceptable toxicity or disease progression as determined by the investigator according to RECIST v1.1.
  Interventions: Drug: Fulvestrant; Drug: Inavolisib; Drug: Atirmociclib

INTERVENTIONS:
Drug: Capecitabine — Capecitabine will be administered 1250 milligrams per square meter (mg/m^2) orally twice daily on Days 1-14 of each 21-day cycle.
  Other Names: RO0091978
  Arms: Capecitabine
Drug: Atezolizumab — For Atezolizumab + SGN-LIV1A, Atezolizumab + Sacituzumab Govitecan, or Atezolizumab + Chemo arms: atezolizumab will be administered intravenously (IV), 1200 mg, on Day 1 of each 21-day cycle.
  For Atezolizumab + Nab-Paclitaxel, Atezolizumab + Selicrelumab + Bevacizumab, Atezolizumab + Ipatasertib, or Atezolizumab + Nab-Paclitaxel + Tocilizumab arms: atezolizumab will be administered IV, 840 mg on Days 1 and 15 of each 28-day cycle.
  Other Names: RO5541267
  Arms: Atezolizumab + Chemo (Gemcitabine + Carboplatin or Eribulin); Atezolizumab + Ipatasertib; Atezolizumab + Nab-Paclitaxel; Atezolizumab + Nab-Paclitaxel + Tocilizumab; Atezolizumab + SGN-LIV1A; Atezolizumab + Sacituzumab Govitecan; Atezolizumab + Selicrelumab + Bevacizumab
Drug: Ipatasertib — Ipatasertib will be administered by mouth 400 mg once a day, on Days 1-21 of each 28-day cycle.
  Arms: Atezolizumab + Ipatasertib
Drug: SGN-LIV1A — SGN-LIV1A will be administered IV, 2.5 milligrams per kilogram (mg/kg) (maximum calculated dose 250 mg), on Day 1 of each 21-day cycle.
  Other Names: RO7235441, Ladiratuzumab vedotin
  Arms: Atezolizumab + SGN-LIV1A
Drug: Bevacizumab — Bevacizumab will be administered IV, 10 mg/kg, on Days 1 and 15 of each 28-day cycle.
  Arms: Atezolizumab + Selicrelumab + Bevacizumab
Drug: Chemotherapy (Gemcitabine + Carboplatin or Eribulin) — Gemcitabine will be administered by IV, 1000 mg/m^2, along with carboplatin, by IV, on Days 1 and 8 of each 21-day cycle.
  Or
  Eribulin will be administered IV, 1.4 mg/m^2 on Days 1 and 8 of each 21-day cycle.
  Arms: Atezolizumab + Chemo (Gemcitabine + Carboplatin or Eribulin)
Drug: Selicrelumab — Selicrelumab will be administered by subcutaneous (SC) injection, at a fixed dose of 16 mg on Day 1 of Cycles 1 to 4 and every third cycle thereafter (Cycle = 28 days).
  Arms: Atezolizumab + Selicrelumab + Bevacizumab
Drug: Tocilizumab — Tocilizumab will be administered IV, 8 mg/kg on Day 1 of each 28-day cycle.
  Other Names: RO4877533
  Arms: Atezolizumab + Nab-Paclitaxel + Tocilizumab
Drug: Nab-Paclitaxel — Nab-Paclitaxel will be administered IV, 100 mg/m^2, on Days 1, 8, and 15 of each 28-day cycle.
  Other Names: RO0247506
  Arms: Atezolizumab + Nab-Paclitaxel; Atezolizumab + Nab-Paclitaxel + Tocilizumab
Drug: Sacituzumab Govitecan — Sacituzumab govitecan will be administered by IV infusion, 10 mg/kg, on Days 1 and 8 of each 21-day cycle.
  Other Names: RO7445735
  Arms: Atezolizumab + Sacituzumab Govitecan
Drug: Abemaciclib — Abemaciclib tablets will be administered at a dose of 150 mg twice daily by mouth on Days 1-28 of each 28-day cycle.
  Other Names: RO7071651
  Arms: Inavolisib + Abemaciclib + Fulvestrant; Inavolisib + Abemaciclib + Letrozole
Drug: Fulvestrant — For Inavolisib + Abemaciclib + Fulvestrant, Inavolisib + Ribociclib (Dose #1) + Fulvestrant, Inavolisib + Ribociclib (Dose #2) + Fulvestrant, or Inavolisib + Atirmociclib + Fulvestrant arms:
  Fulvestrant 500 mg, administered as an IM injection on Days 1 and 15 of Cycle 1, followed by Day 1 of each 28-day cycle thereafter.
  For Empa + Inavolisib + Fulvestrant ± Palbociclib, or Metformin + Inavolisib + Fulvestrant ± Palbociclib arms:
  Fulvestrant 500 mg, administered as an IM injection on Day 1 and as per local prescribing guidelines thereafter.
  Arms: Empagliflozin (Empa) + Inavolisib (Inavo) + Fulvestrant (Fulv) ± Palbociclib (Palbo); Inavolisib + Abemaciclib + Fulvestrant; Inavolisib + Atirmociclib (Atirmo) + Fulvestrant; Inavolisib + Ribociclib (Dose #1) + Fulvestrant; Inavolisib + Ribociclib (Dose #2) + Fulvestrant; Metformin (Metf) + Inavolisib + Fulvestrant ± Palbociclib
Drug: Ribociclib (Dose #1) — Ribociclib tablets will be administered by mouth once daily.
  Other Names: RO7072612
  Arms: Inavolisib + Ribociclib (Dose #1) + Fulvestrant; Inavolisib + Ribociclib (Dose #1) + Letrozole
Drug: Inavolisib (Dose #1) — Inavolisib tablets will be administered by mouth once daily.
  Other Names: GDC-0077, RO7113755
  Arms: Inavolisib (Dose #1) + Trastuzumab Deruxtecan
Drug: Trastuzumab Deruxtecan — Trastuzumab Deruxtecan will be administered IV, 5.4 mg/kg on Day 1 of each 21-day cycle.
  Arms: Inavolisib (Dose #1) + Trastuzumab Deruxtecan; Inavolisib (Dose #2) + Trastuzumab Deruxtecan
Drug: Ribociclib (Dose #2) — Ribociclib tablets will be administered by mouth once daily.
  Other Names: RO7072612
  Arms: Inavolisib + Ribociclib (Dose #2) + Fulvestrant; Inavolisib + Ribociclib (Dose #2) + Letrozole
Drug: Letrozole — Letrozole tablets will be administered at a dose of 2.5 mg once a day by mouth on Days 1-28 of each 28-day cycle.
  Arms: Inavolisib + Abemaciclib + Letrozole; Inavolisib + Ribociclib (Dose #1) + Letrozole; Inavolisib + Ribociclib (Dose #2) + Letrozole
Drug: Inavolisib (Dose #2) — Inavolisib tablets will be administered by mouth once daily.
  Other Names: GDC-0077, RO7113755
  Arms: Inavolisib (Dose #2) + Trastuzumab Deruxtecan
Drug: Inavolisib — Inavolisib tablets will be administered by mouth OD.
  Other Names: GDC-0077, RO7113755
  Arms: Empagliflozin (Empa) + Inavolisib (Inavo) + Fulvestrant (Fulv) ± Palbociclib (Palbo); Inavolisib + Abemaciclib + Fulvestrant; Inavolisib + Abemaciclib + Letrozole; Inavolisib + Atirmociclib (Atirmo) + Fulvestrant; Inavolisib + Ribociclib (Dose #1) + Fulvestrant; Inavolisib + Ribociclib (Dose #1) + Letrozole; Inavolisib + Ribociclib (Dose #2) + Fulvestrant; Inavolisib + Ribociclib (Dose #2) + Letrozole; Metformin (Metf) + Inavolisib + Fulvestrant ± Palbociclib
Drug: Empagliflozin — Empagliflozin, administered orally, once daily (QD)
  Arms: Empagliflozin (Empa) + Inavolisib (Inavo) + Fulvestrant (Fulv) ± Palbociclib (Palbo)
Drug: Palbociclib — For Empagliflozin + Inavolisib + Fulvestrant ± Palbociclib arm:
  Palbociclib 125 mg administered orally, QD in Cycle 1 followed by 125 mg on Days 1-21 of each cycle.
  For Metformin + Inavolisib + Fulvestrant ± Palbociclib arm: Palbociclib 125 mg administered orally, QD in Cycle 1, followed by 125 mg on Days 1-21 of each cycle (Cycle=28 days).
  Arms: Empagliflozin (Empa) + Inavolisib (Inavo) + Fulvestrant (Fulv) ± Palbociclib (Palbo); Metformin (Metf) + Inavolisib + Fulvestrant ± Palbociclib
Drug: Metformin — Metf 1000 mg administered orally QD.
  Arms: Metformin (Metf) + Inavolisib + Fulvestrant ± Palbociclib
Drug: Atirmociclib — Atirmociclib administered orally, BID on Days 1-28 for each 28-day cycle.
  Arms: Inavolisib + Atirmociclib (Atirmo) + Fulvestrant

SUMMARY:
This is an umbrella study evaluating the efficacy and safety of multiple treatment combinations in participants with metastatic or inoperable locally advanced breast cancer.

The study will be performed in two stages. During Stage 1, six cohorts will be enrolled in parallel in this study:

Cohort 1 will consist of programmed death-ligand 1 (PD-L1)-positive participants who have received no prior systemic therapy for metastatic or inoperable locally advanced triple-negative breast cancer (TNBC) (first-line [1L] PD-L1+ cohort).

Cohort 2 will consist of participants who had disease progression during or following 1L treatment with chemotherapy for metastatic or inoperable locally-advanced TNBC and have not received cancer immunotherapy (CIT) (second-line [2L] CIT-naïve cohort).

Cohort 3, 5, and 6 will consist of participants with locally advanced or metastatic hormone receptor-positive (HR+), human epidermal growth factor receptor 2 (HER2)-negative disease with one or more PIK3CA mutations.

Cohort 4 will consist of participants with locally advanced or metastatic HER2+ /HER2-low disease with one or more PIK3CA mutations who had disease progression on standard-of-care therapies (HER2+ /HER2-low cohort).

In each cohort, eligible participants will initially be assigned to one of several treatment arms (Stage 1). During Stage 2, participants in the 2L CIT-naïve cohort who experience disease progression, loss of clinical benefit, or unacceptable toxicity during Stage 1 may be eligible to continue treatment with a different treatment combination, provided Stage 2 is open for enrollment and all eligibility criteria are met.

ELIGIBILITY:
Inclusion Criteria

Patients must meet all of the following criteria to qualify for Stage 1 (all cohorts) and to qualify for Stage 2 (2L CIT-naïve cohort):

* Age >/= 18 years at the time of signing Informed Consent Form
* Eastern cooperative oncology group (ECOG) performance status of 0 or 1
* Able to comply with the study protocol, in the investigator's judgment
* Metastatic or inoperable locally advanced breast cancer
* Measurable disease (at least one target lesion) according to RECIST v1.1
* Life expectancy >/= 3 months, as determined by the investigator
* Tumor accessible for biopsy, unless archival tissue is available
* Availability of a representative tumor specimen that is suitable for biomarker analysis via central testing
* Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from breastfeeding and donating eggs, as outlined for each specific treatment arm
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as outlined for each specific treatment arm

Exclusion Criteria

Exclusion Criteria for Stage 1

* Prior treatment with T-cell co-stimulating or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies, CD40 agonists or interleukin-2 (IL-2) or IL-2-like compounds
* Biologic treatment (e.g., bevacizumab) within 2 weeks prior to initiation of study treatment, or other systemic treatment for TNBC within 2 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor alpha agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during the course of the study
* Eligibility only for the control arm

Exclusion Criteria for Stage 1 (both cohorts) and Stage 2 (2L CIT-naïve cohort)

* Adverse events from prior anti-cancer therapy that have not resolved to Grade </= 1 or better with the exception of alopecia of any grade and Grade </= 2 peripheral neuropathy
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)
* Uncontrolled tumor-related pain
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* History of leptomeningeal disease
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Active tuberculosis
* Severe infection within 4 weeks prior to initiation of study treatment
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment
* Significant cardiovascular disease
* Prior allogeneic stem cell or solid organ transplantation
* History of malignancy other than breast cancer within 2 years prior to screening, with the exception of those with a negligible risk of metastasis or death
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 792 (Estimated)
Dates: Start 2018-03-30 (Actual); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Baseline until disease progression or loss of clinical benefit (up to approximately 10 years)

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the end of study (up to approximately 10 years) as determined by the investigator according to RECIST v1.1
Disease Control Rate (DCR) | Baseline through end of study (up to approximately 10 years)
Overall Survival (OS) | Randomization to death from any cause, through the end of study (up to approximately 10 years)
Overall Survival (at specific time-points) | 12 and 18 months
Duration of Response (DOR) | Randomization until first occurrence of a documented objective response to the first recorded occurrence of disease progression or death from any cause (whichever occurs first), through end of study (up to approximately 10 years)
Percentage of Participants with Adverse Events | Baseline to end of study (up to approximately 10 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (45):
- United States (16):
  - City of Hope, Duarte, California
  - University of California San Diego Medical Center, La Jolla, California
  - Stanford Cancer Institute, Stanford, California
  - Rocky Mountain Cancer Center - Longmont, Longmont, Colorado
  - H. Lee Moffitt Cancer Center and Research Inst., Tampa, Florida
  - Hackensack Univ Medical Center, Hackensack, New Jersey
  - Regional Cancer Care Associates, LLC, Howell Township, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYU Langone Medical Center, New York, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Tennessee Oncology - Chattanooga Oncology & Hematology Associates, Chattanooga, Tennessee
  - The West Clinic, Germantown, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology-Plano East, Plano, Texas
- Australia (2):
  - Peter MacCallum Cancer Centre-East Melbourne, Melbourne, Victoria
  - Fiona Stanley Hospital - Medical Oncology, Murdoch, Western Australia
- France (4):
  - Centre Léon Bérard, Lyon
  - Institut régional du Cancer Montpellier, Montpellier
  - Institut Universitaire du Cancer de Toulouse-Oncopole, Toulouse
  - Gustave Roussy, Villejuif
- Germany (2):
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
- Israel (7):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Medical Center, Jerusalem
  - Rabin MC, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Assuta Medical Centers, Tel Aviv
- South Korea (5):
  - National Cancer Center Clinical Trials Center / Center for Breast Cancer, Goyang-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - University of Ulsan College of Medicine - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Hospital del Mar, Barcelona
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Centro Integral Oncológico Clara Campal Ensayos Clínicos START, Madrid
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- United Kingdom (2):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Barts Health NHS Trust - St Bartholomew's Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing